CLINICAL TRIAL: NCT03457129
Title: Fycompa Titration Intervals and Effects on Retention Rate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Principal Investigator, Stephanie Marsh, Clinical Research Coordinator, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fycompa Titration IIS
Record Dates: First submitted 2017-11-03; First posted 2018-03-07 (Actual); Results first posted 2021-12-08 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; Epilepsy, partial onset; Epilepsy, generalized onset; Fycompa; perampanel
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fycompa 2 week titration intervals (Active Comparator): Perampanel oral tablet: 2mg by mouth every 24 hours for two weeks, then up-titrated by 2 mg every two weeks to a target dose of 6 mg/day. Minimum total daily dose = 2 mg/day. Maximum daily dose is 12 mg/day. Total daily dose will be determined by the Investigator based on tolerability and seizure control.
  Interventions: Drug: Perampanel Oral Tablet
- Fycompa 3 week titration intervals (Experimental): Perampanel oral tablet: 2mg by mouth every 24 hours for three weeks, then up-titrated by 2 mg every three weeks to a target dose of 6 mg/day. Minimum total daily dose = 2 mg/day. Maximum daily dose is 12 mg/day. Total daily dose will be determined by the Investigator based on tolerability and seizure control.
  Interventions: Drug: Perampanel Oral Tablet

INTERVENTIONS:
Drug: Perampanel Oral Tablet — Perampanel is an AMPA receptor blockade, that has shown to be efficacious for seizure reduction in both partial onset seizures and generalized tonic-clonic seizures. Perampanel was approved by the FDA in October 2012 as adjunctive treatment in patients with partial onset seizures. Additionally, in June 2015, Fycompa was approved as adjunctive therapy in patients with primary generalized tonic clonic seizures.
  Other Names: Fycompa

SUMMARY:
This study will aim to improve retention and tolerability by slowing the initial titration rate of perampanel from a standard up-titration rate of 2 week intervals to a slower up-titration rate consisting of 3 week intervals. Subjects will be randomized to either perampanel, standard titration interval rate (Group A) or perampanel, slower titration interval rate (Group B).

DETAILED DESCRIPTION:
A total of 60 subjects with a confirmed diagnosis of either partial onset or primary generalized epilepsy will be recruited into the trial. 30 subjects will initiate perampanel at a dose of 2 mg/day and titrate upwards every 2 weeks to a target dose of 6 mg/day. Subjects in this group will be designated Group A. The remaining 30 subjects will also begin perampanel at a dose of 2 mg/day but will titrate upwards every 3 weeks to a target dose of 6 mg/day and will be designated Group B.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide written informed consent signed by the subject or legal guardian prior to entering the study in accordance with ICH and GCP guidelines.
2. Subject has a confirmed diagnosis of medically refractory epilepsy with or without secondary generalization for at least 12 months prior to visit 1.
3. Subjects currently being treated with 1 to 3 antiepileptic medications with or without VNS (does not count as an AED).
4. Subjects aged 18 to 75.
5. Subject's requiring an additional epilepsy medication due to either uncontrolled seizures and/or lack of tolerability with current epilepsy medications.
6. Can be safely treated, in the opinion of the investigator, with Fycompa.
7. Able and agrees to follow the specified titration schedule.
8. Subjects or a legal guardian who is able to communicate effectively with study personnel and considered reliable, able, willing and cooperative with regard to complying with protocol-defined requirements, including completion of the study diary.

Exclusion Criteria:

1. Any history of non-epileptic or psychogenic seizures.
2. Women who are currently pregnant, lactating or have plans to become pregnant in the immediate future.
3. Subjects with active suicidal ideation or behavior as evidenced by positive answers on the Columbia Suicide Severity Rating Scale (C-SSRS) or subject's with a history of suicidal ideation or attempt within 12 months.
4. Subjects with a suicidal attempt in the 12 months prior to Visit 1
5. Any clinically significant medical or psychiatric illness, psychological or behavioral problems, which in the opinion of the investigator would interfere with the subject's ability to participate in the study.
6. Subjects with severe hepatic impairment or severe renal impairment or on hemodialysis.
7. Any use of concomitant medication as listed in the drug insert, including medications known to be inducers of cytochrome P450 (CYP3A).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman C Wang, MD, Principal Investigator — Banner University Medical Center
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data with other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fycompa 2 Week Titration Intervals | Fycompa 3 Week Titration Intervals
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fycompa 2 Week Titration Intervals | Fycompa 3 Week Titration Intervals | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (11) | 43 (9) | 37 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 10 | 18
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Completing 52 Weeks of Adjunctive Therapy During the Maintenance Phase [Retention Rate].
Description: Retention rate, which indirectly measures the therapeutic tolerance, will be measured at 52 weeks in each group.
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Fycompa 2 Week Titration Intervals | Fycompa 3 Week Titration Intervals
Number analyzed (Participants) | 7 | 8
Participants | 2 | 3

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events (TEAEs) Reported by the Subject or Observed by the Investigator [Safety and Tolerability].
Description: Adverse events experienced in each group will be tabulated and the total percentage of subjects reporting adverse events will be calculated.
Time Frame: Up to 52 weeks
Measure: Number; unit: participants
Arm/Group | Fycompa 2 Week Titration Intervals | Fycompa 3 Week Titration Intervals
Number analyzed (Participants) | 10 | 10
participants | 4 | 3

3. Secondary Outcome: Seizures Frequency Per Week
Description: The average of seizures per week will be calculated starting at initial titration through final maintenance [Efficacy]."
Time Frame: Up to 52 weeks
Population: 2 participants in Group A were discontinued due to adverse events and 3 were lost to follow-up. In group B, 3 participants were discontinued due to adverse events and 2 were lost to follow-up. Therefore, only 5 participants remained in each treatment group for determination of seizure frequency during the final maintenance phase.
Measure: Mean (Standard Deviation); unit: Seizures per week
Arm/Group | Fycompa 2 Week Titration Intervals | Fycompa 3 Week Titration Intervals
Number analyzed (Participants) | 5 | 5
Seizures per week | 0.912 (0.647) | 0.508 (0.887)

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Arm/Group | Fycompa 2 Week Titration Intervals | Fycompa 3 Week Titration Intervals
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10
Other Adverse Events (participants affected / at risk) | 4/10 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fycompa 2 Week Titration Intervals (N=10) | Fycompa 3 Week Titration Intervals (N=10)
Intractable Seizures (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fycompa 2 Week Titration Intervals (N=10) | Fycompa 3 Week Titration Intervals (N=10)
Anger (Psychiatric disorders) | 4 | 3
Drowsiness (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Numbness (Nervous system disorders) | 0 | 1
Unsteadiness (Nervous system disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 1
Memory difficulty (Nervous system disorders) | 0 | 1
Anxiety (Nervous system disorders) | 1 | 0
Abnormal menses (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Speech difficulty (Nervous system disorders) | 1 | 0
Sleep difficulty (Nervous system disorders) | 1 | 1
Head cold (Infections and infestations) | 1 (1) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT03457129/Prot_SAP_000.pdf